CLINICAL TRIAL: NCT03245281
Title: LINQ for impEdance meAsuremeNt While Off From HF Medication Study
Acronym: LEAN HF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MDT16014
Record Dates: First submitted 2017-07-07; First posted 2017-08-10 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Diuretics

STUDY DESIGN:
Intervention Model Description: According to the enrolment chronological order, each subject will be allocated to Diuretic Suspension group (DS), Diuretic Increase (DI) or Diuretic+MRA medication Suspension (DMS), which will define the medication regimen before the follow-up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diuretic Suspension (DS) (Experimental)
  Interventions: Drug: Diuretic Suspension (DS)
- Diuretic Increase (DI) (Experimental)
  Interventions: Drug: Diuretic Increase (DI)
- Diuretic and Medication Suspension (DMS) (Experimental)
  Interventions: Drug: Diuretic and Medication Suspension (DMS)

INTERVENTIONS:
Drug: Diuretic Suspension (DS) — Stop diuretic consumption in the 48h before the follow-up visit
  Arms: Diuretic Suspension (DS)
Drug: Diuretic Increase (DI) — Double diuretics dosage in the 48h before the follow-up visit
  Arms: Diuretic Increase (DI)
Drug: Diuretic and Medication Suspension (DMS) — Stop diuretic and MRA medication consumption in the 48h before the follow-up visit
  Arms: Diuretic and Medication Suspension (DMS)

SUMMARY:
The purpose of this non-randomized, cross-over, unblinded, single-center feasibility study is to assess the sensitivity of the LINQ ICM to measure derived-subcutaneous impedance in patients with heart failure during periods when diuretics and/or HF-medication consumption is increased or suspended for 48 hours (up to 72 hours at physician discretion) and to collect safety information related to HF status and to medication consumption changes.

DETAILED DESCRIPTION:
Up to 30 subjects with a clinical diagnosis of Heart Failure will be enrolled in the study. It is expected that the subjects will be enrolled over a period of approximately 6 months.

3 follow up visits are planned at 2, 4 and 6 months (+/- one week) following the LINQ ICM implant.

The total expected duration of the study is of about 1 year. According to the enrolment chronological order, each subject will be allocated to Diuretic Suspension group (DS), Diuretic Increase (DI) or Diuretic+MRA medication Suspension (DMS), which will define the medication regimen before the follow-up visit.

Primary objective of the study is detecting the variation of impedance magnitude and the time of occurrence after medication regimen changes will be evaluated at each follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Heart Failure
* Plasma NT-proBNP (>250ng/L in SR and >1,000ng/L in AF)
* LVEF <50% measured in the year before enrolment
* Treated routinely with a daily dose of loop diuretic
* Receiving other guideline-indicated therapy for heart failure
* Willing to sign the informed consent form.
* Greater than 18 years of age.

Exclusion Criteria:

* Pregnant patients (all females of child-bearing potential must have a negative pregnancy test before LINQ ICM implant)
* eGFR <30 ml/minute.
* Any concomitant condition which in the opinion of the investigator would not allow a safe participation in the study.
* Patients with implanted pacemakers or defibrillators
* Severe aortic or mitral valve disease
* Breathlessness at rest or on minor exertion.
* Chest pain at rest or on mild or moderate exertion.
* Patients deemed too unstable to miss 48 hours of heart failure treatment
* Enrolled in another study that could confound the results of this study, without documented pre-approval from Medtronic study manager

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Derived-subcutaneous impedance | 2 months
  The variation of impedance magnitude and the time of occurrence after medication regimen changes will be detected by the LINQ ICM

SECONDARY OUTCOMES:
Number of Adverse Events | 6 months
  All AEs related to changes in the therapeutic regimen and/or to HF status will be collected through CRF completion
Number of Transitory Arrhythmias | 6 months
  Any transitory arrhythmias related to drug regimen changes and/or HF condition will be collected through CRF completion

CONTACTS AND LOCATIONS:
Overall Officials: John Cleland, Prof, Study Chair — NHS Greater Glasgow & Clyde
Locations (1):
- Nhs Greater Glasgow & Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Butler J, Arbogast PG, Daugherty J, Jain MK, Ray WA, Griffin MR. Outpatient utilization of angiotensin-converting enzyme inhibitors among heart failure patients after hospital discharge. J Am Coll Cardiol. 2004 Jun 2;43(11):2036-43. doi: 10.1016/j.jacc.2004.01.041. PMID 15172409
- [Background] Monane M, Bohn RL, Gurwitz JH, Glynn RJ, Avorn J. Noncompliance with congestive heart failure therapy in the elderly. Arch Intern Med. 1994 Feb 28;154(4):433-7. PMID 8117176
- [Background] Mittal S, Sanders P, Pokushalov E, Dekker L, Kereiakes D, Schloss EJ, Pouliot E, Franco N, Zhong Y, DI Bacco M, Purerfellner H. Safety Profile of a Miniaturized Insertable Cardiac Monitor: Results from Two Prospective Trials. Pacing Clin Electrophysiol. 2015 Dec;38(12):1464-9. doi: 10.1111/pace.12752. Epub 2015 Oct 20. PMID 26412309
- [Background] Purerfellner H, Sanders P, Pokushalov E, Di Bacco M, Bergemann T, Dekker LR; Reveal LINQ Usability Study Investigators. Miniaturized Reveal LINQ insertable cardiac monitoring system: First-in-human experience. Heart Rhythm. 2015 Jun;12(6):1113-9. doi: 10.1016/j.hrthm.2015.02.030. Epub 2015 Feb 26. PMID 25728756
- [Background] van der Wal MH, Jaarsma T, van Veldhuisen DJ. Non-compliance in patients with heart failure; how can we manage it? Eur J Heart Fail. 2005 Jan;7(1):5-17. doi: 10.1016/j.ejheart.2004.04.007. PMID 15642526